CLINICAL TRIAL: NCT00000334
Title: Pharmacological Comparison of Buprenorphine and Methadone
Brief Title: Comparison of Buprenorphine and Methadone - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-3-0009-3; Y01-3-0009-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare agonist and antagonist profile associated with buprenorphine vs. methadone during opiate withdrawal.

ELIGIBILITY:
Please contact site for information.

Ages: 23 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 2002-12-01 (Actual); Primary Completion 2004-11-01 (Actual); Study Completion 2005-01-15 (Actual)

PRIMARY OUTCOMES:
Withdrawal severity
Opiate agonist symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deutsch, M.D., Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC VA, Washington D.C., District of Columbia, United States